CLINICAL TRIAL: NCT02692313
Title: Hypoglycemia Associated Autonomic Dysfunction Dose Response of Epinephrine
Brief Title: Dose Response of Epinephrine
Acronym: Epineprhine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Stephen N. Davis, MBBS, Chairman of Medicine, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00068487
Record Dates: First submitted 2016-02-10; First posted 2016-02-26 (Estimated); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Complications
Keywords: epinephrine; counterregulation; dose responses
MeSH Terms: conditions — Diabetes Complications | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Saline infusion (Placebo Comparator): Hyperinsulinemic euglycemic glucose clamp with saline infusion
  Interventions: Other: Saline infusion
- Epinephrine infusion-0.015ug/kg/min (Experimental): Hyperinsulinemic euglycemic glucose clamp with epinephrine infusion of 0.015 ug/kg/min
  Interventions: Drug: Epinephrine
- Epinephrine infusion-0.03 ug/kg/min (Experimental): Hyperinsulinemic euglycemic glucose clamp with epinephrine infusion of 0.03 ug/kg/min
  Interventions: Drug: Epinephrine
- Epinephrine infusion-0.06 ug/kg/min (Experimental): Hyperinsulinemic euglycemic glucose clamp with epinephrine infusion of 0.06 ug/kg/min
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Epinephrine — Dose response of epinephrine infusion
  Other Names: Adrenaline
  Arms: Epinephrine infusion-0.015ug/kg/min; Epinephrine infusion-0.03 ug/kg/min; Epinephrine infusion-0.06 ug/kg/min
Other: Saline infusion — Placebo
  Other Names: Placebo
  Arms: Saline infusion

SUMMARY:
Epinephrine is the principal physiologic defense against hypoglycemia in type 1 and longer duration type 2 DM. Despite this, it is unknown how epinephrine regulates in-vivo endothelial function and atherothrombotic balance in humans. The specific aim of our study will be to determine the dose response effects of the key ANS counterregulatory hormone epinephrine on endothelial function, fibrinolytic balance and pro-atherogenic inflammatory mechanisms in healthy humans.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls age 18-55 yr.
* Body mass index >21 kg · m-2

Exclusion Criteria:

* Pregnant or breastfeeding women
* Subjects unwilling or unable to comply with approved contraception measures
* Subjects unable to give voluntary informed consent
* Subjects on anticoagulant drugs, anemic or with known bleeding diatheses
* Subjects with a history of severe, uncontrolled hypertension, heart disease, cerebrovascular incidents
* Current tobacco use
* Subjects with any known allergies to any of the study medications being used

Physical Exam Exclusion Criteria

* Uncontrolled severe hypertension (i.e., blood pressure greater than 160/100)
* Clinically significant cardiac abnormalities (e.g. heart failure, arrhythmia)
* Pneumonia treatment or hospitalization within 2 weeks prior to enrollment (study visit)
* Hepatic failure / jaundice
* Renal failure
* Cerebrovascular accident occurrence or hospitalization within 4 weeks prior to enrollment
* Fever greater than 38.0 degrees C

Screening Laboratory Tests Exclusion Criteria

* Hematocrit lower than 32 %
* White blood cell (WBC) count lower than 3 thou/ul or greater than 14 thou/ul
* Liver function tests: serum glutamic oxaloacetic transaminase (SGOT) and serum glutamic-pyruvic transaminase (SGPT) greater than twice upper limit of normal range
* Alkaline phosphatase greater than 150U/L
* Total bilirubin (TBil) greater than 2 mg/dl
* Estimated glomerular filtration rate (eGFR) less than 60 mL/min/1.73 m2
* Positive human immunodeficiency virus (HIV), Hepatitis B or Hepatitis C
* Any abnormal cardiac response during multi-stage exercise test (if over 40 years of age)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-06; Primary Completion 2025-09 (Actual); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation (FMD) of the brachial artery | From baseline (pre glucose clamp) to end of experiment (time 240 minutes- 2 hours post intervention (glucose clamp))
  Measurements of FMD will be taken at baseline (pre intervention) and end of glucose clamp (post intervention) and the maximal % change determined

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Davis, MBBS, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland, Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No